CLINICAL TRIAL: NCT06365762
Title: A Phase 1/2, Randomized, Placebo-Controlled, Double-Masked, Multicenter, Dose-Ranging, Safety and Efficacy of C-KAD Ophthalmic Solution in Patients With Loss of Contrast Sensitivity Due to Age-Related, Low-Grade Nuclear Cataract
Brief Title: The Safety and Efficacy Study of Ethylenediaminetetraacetic Acid (EDTA) Ophthalmic Solution in Patients With Loss of Contrast Sensitivity Due to Age-Related, Low-Grade Nuclear Cataract
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Livionex Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CK-0103
Record Dates: First submitted 2024-04-10; First posted 2024-04-15 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2024-04

CONDITIONS: Age Related Cataracts
Keywords: Contrast Sensitivity
MeSH Terms: interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- C-KAD 2.6% (Experimental): Administered four times a day (QID; no less than 3 hours apart) in both eyes for 120 days
  Interventions: Drug: EDTA Ophthalmic Solution 2.6%
- C-KAD 1.3% (Experimental): Administered four times a day (QID; no less than 3 hours apart) in both eyes for 120 days
  Interventions: Drug: EDTA Ophthalmic Solution 1.3%
- Placebo (Placebo Comparator): Administered four times a day (QID; no less than 3 hours apart) in both eyes for 120 days
  Interventions: Drug: Saline Solution (Placebo)

INTERVENTIONS:
Drug: EDTA Ophthalmic Solution 2.6%
  Other Names: C-KAD 2.6%
  Arms: C-KAD 2.6%
Drug: EDTA Ophthalmic Solution 1.3%
  Other Names: C-KAD 1.3%
  Arms: C-KAD 1.3%
Drug: Saline Solution (Placebo)
  Other Names: Software Saline
  Arms: Placebo

SUMMARY:
The study objectives were:

* To evaluate the efficacy of EDTA 1.3% and 2.6% ophthalmic solution (C-KAD) in improving visual function as assessed by contrast sensitivity;
* To evaluate the safety and tolerability of two doses of EDTA ophthalmic solution (C-KAD); and
* To determine the optimal clinical dose of EDTA ophthalmic solution (C-KAD) which to proceed into pivotal study(s).

DETAILED DESCRIPTION:
This was a prospective, randomized, placebo-controlled, double-masked, parallel evaluation of the safety and efficacy of EDTA ophthalmic solution in patients with loss of contrast sensitivity due to age-related, low-grade cataract.

111 subjects were enrolled at six study sites within the U.S. and randomly assigned in 1:1:1 ratio to treatment with 2.6% C-KAD, 1.3% C-KAD and placebo. The treatment duration was 120 days with a run-in period and follow-up period of 14 days each.

During the Run-in Period, patients received pre-treatment with lubricating eye drops (Refresh® Plus Lubricant Eye Drops) in both eyes to ensure uniformity in the level of ocular hydration at Baseline in patients randomized into the study.

Patients were evaluated at a Screening Visit (Day -14), at Baseline (Day 0), during the dosing period (Days 30, 60, 90, 120) and at the Follow-up Visit (Day 134), two weeks after completion of active treatment.

Tolerability and efficacy were assessed by Slit Lamp and Fundus Examinations, Best-Corrected Distance Visual Acuity, Contrast Sensitivity, Endothelial Cell Count, Pentacam Imaging, Tear Film Break-Up Time, IOP measurements, Pupil Size measurement and evaluation of Adverse Events.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients ≥ 50 years of age
* Presence of early nuclear sclerosis cataract in both eyes below the level recommended for surgical replacement
* Both eyes having contrast sensitivity measurements of:

  * Screening Visit:
  * Less than or equal to 6, 4 and 4 in spatial frequencies C, D and E, respectively under mesopic illumination
  * Baseline Visit:
  * Less than or equal to 6, 4 and 4 in spatial frequencies C, D and E, respectively under mesopic illumination and
  * Greater than 0 in all five spatial frequencies (Patches A, B, C, D and E) under photopic illumination
* Best-Corrected Distance Visual Acuity (BCDVA) measurement by ETDRS of better than or equal to 20/50 in both eyes attributable to low- grade nuclear cataract
* Patient must be willing and able to provide written informed consent
* Patient must be willing and able to comply with study visits as described in the protocol

Exclusion Criteria:

* Clinical evidence of any active ocular infection (i.e., bacterial, viral, parasitic or fungal) in either eye
* History of herpetic ocular infection in either eye
* Presence or history of glaucoma in either eye
* Presence or history of intraocular pressure of >22 mm Hg in either eye
* Amblyopia in either eye
* Presence of any corneal disorder including pterygium or superficial keratitis
* Dry eyes which require the use of a prescription medication
* Presence of posterior subcapsular cataract
* Presence of cortical cataract that intrudes within the central 4mm of the lens
* Presence or history of any ocular inflammatory disorder in either eye (e.g., uveitis, ocular allergies)
* Patients with known allergies to EDTA preservatives
* Presence of any optic nerve or retinal disorders including, but not limited to, age-related macular degeneration, optic neuropathy, etc. in either eye
* Prior intraocular, refractive and/or laser surgery of any type in either eye
* Anticipated need for ocular surgery in either eye within six months of study enrollment
* History of diabetes
* Pseudo-exfoliation syndrome
* Contact lens use (soft contact lens wear within 2 weeks of the date of randomization, rigid lens wear within three months of the date of randomization. No contact lens use throughout duration of the study)
* Current use or anticipated use of any ocular medications (over-the- counter or prescription). Use of topical ophthalmic drugs should be discontinued 14 days prior to enrollment into the treatment arm of the study
* Current or anticipated use of any systemic or ocular steroids or chronic use of topical steroids within 30 days of study enrollment
* Females who are pregnant, lactating or pre- or peri menopausal and unwilling to use adequate birth control for the duration of the study
* Participation in an investigational device or drug trial within the last 30 day
* Presence of any condition, abnormality or situation at Screening or at Baseline that in the opinion of the Principal Investigator may preclude the patient's ability to comply with study requirements, including completion of the study or the quality of the data

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 111 (Actual)
Dates: Start 2006-01-01 (Actual); Primary Completion 2006-12-31 (Actual); Study Completion 2007-04-30 (Actual)

PRIMARY OUTCOMES:
Contrast Sensitivity (Mesopic) Responder Analysis | Baseline, Days 30, 60, 90, and 120
  Proportion of patients with ≥ 2-patch (0.30 logCS) contrast sensitivity improvement in at least two spatial frequencies under mesopic illumination

SECONDARY OUTCOMES:
Cumulative Improvement in Contrast Sensitivity (Mesopic) | Baseline, Days 30, 60, 90, and 120
  total changes in patches of contrast sensitivity measurements across all five spatial frequencies (1.5, 3, 6, 12, and 18 cycles per degree)

OTHER OUTCOMES:
Mean Change in Contrast Sensitivity (Mesopic) | Baseline, Days 30, 60, 90, and 120
  Mean change in contrast sensitivity from baseline under mesopic illumination
Mean Change in Best-Corrected Visual Acuity (BCVA) | Baseline, Days 30, 60, 90, and 120
  Mean change in BCVA from baseline using ETDRS charts
Pentacam Imaging | Baseline, Baseline, Days 120
  Densitometric Analysis using Scheimpflug Images (substudy patients at a selected study site only)

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - St Mary's Eye Specialists, Inc., San Francisco, California
  - Hunkeler Eye Institute, Overland Park, Kansas
  - The Johns Hopkins Hospital & Health System, Wilmer Eye Institute, Lutherville, Maryland
  - Harvard Medical School, Massachusetts Eye and Ear Infirmary, Boston, Massachusetts
  - Charlotte Eye, Ear, Nose, and Throat Associates, Charlotte, North Carolina
  - University of Utah, John Moran Eye Center, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No